CLINICAL TRIAL: NCT05390931
Title: The Effect of Motivational Interviews on Cardiovascular Disease Risks and Healthy Lifestyle Behavior Changes in Essential Hypertension Patients: A Randomized Controlled Study
Brief Title: Effect of Motivational Interviews on Cardiovascular Disease Risks and Healthy Lifestyle Behavior Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, Assistant Professor Doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FirdesKomaç
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Essential Hypertension; Motivational Interview; Cardiovascular Disease Risk; Healthy Lifestyle Behavior
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the study, participants will be left unaware of whether they are in the study or control group (single-blind masking).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group intervention consists of 6-session motivational interviews (6 times in total, once every month), a health education structured according to the health belief model, a training booklet on healthy lifestyle behavior changes at the end of the training, and 6-month follow-up.
  Interventions: Behavioral: 6-session motivational interviews; Other: Health education structured according to the health belief model; Other: Training booklet prepared by the researchers on healthy lifestyle behavior changes; Other: 6 month follow-up
- Control group (Other): Control group intervention consists of a health education structured according to the health belief model, a training booklet on healthy lifestyle behavior changes at the end of the training, and a 6-month follow-up.
  Interventions: Other: Health education structured according to the health belief model; Other: Training booklet prepared by the researchers on healthy lifestyle behavior changes; Other: 6 month follow-up

INTERVENTIONS:
Behavioral: 6-session motivational interviews — A total of 6 motivational interviews will be held once a month. Motivational interviews will be conducted individually.
  Arms: Study group
Other: Health education structured according to the health belief model — After the participants enrolled in the study, the patients in the study group will be given a health education structured according to the health belief model at the first interview.
Other: Training booklet prepared by the researchers on healthy lifestyle behavior changes — After the participants enrolled in the study and take health education, a training booklet prepared by the researchers on healthy lifestyle behavior changes will be given to the participants.
Other: 6 month follow-up — Follow-ups will be made 3 times in total, on the basis of pre-test, intermediate follow-up test (3 months), and post-test (6 months).

SUMMARY:
The primary aim of this study is to determine the effects of education and motivational interviews structured according to the health belief model on cardiovascular disease risks and healthy lifestyle behavior changes in patients with an essential hypertension diagnosis. The secondary aim of the study is to determine the effects of the variables that mediate the probability of performing primary prevention measures according to the health belief model of patients with a diagnosis of essential hypertension. The study was planned in a single-center, single-blind, one-to-one, parallel-group, randomized controlled trial design with a 6-month follow-up period. The research will be carried out at Işıklar Family Health Center located in Eskişehir city center in Turkey. The study population of this research consists of 659 patients with a diagnosis of essential hypertension, aged between 30-59 years, registered in Işıklar Family Health Center. The number of samples required for the study was determined by the power analysis made in the GPower 3.1 package program. Assuming that there may be losses during the follow-up and considering the possibility of nonparametric testing, a total of 80 individuals, 40 in each group, with an increase of 20%, will form the research group. The research data collection process will be carried out in 4 stages. First of all, the data required to query the inclusion criteria and exclusion criteria for participant admission to the study will be evaluated using the "Data form for participant admission". For the other stages of the research data collection process; "Pre-test (Beginning at 0 months)", "Intermediate follow-up test (Follow-up at 3 months)" and "Posttest (6 months)" will be administered to the participants in the study and control groups by the researcher. In this study, "Cardiovascular Disease Risk Awareness Assessment Scale", "Cardiovascular Diseases Risk Factors Knowledge Level", "Framingham Cardiovascular Risk Score", "Healthy Lifestyle Behaviors Scale-II", "Hypertension Self-Care Profile", "Hill- Bone Hypertension Treatment Adherence Scale", "Physical Activity Questionnaire for Primary Care" and "SF-12 Quality of Life Scale" will be used as data collection tools. In addition to their routine care, the control group will be given a health education structured according to the health belief model and a training booklet on healthy lifestyle behavior changes at the end of the training.

DETAILED DESCRIPTION:
Hypertension plays an important role in the early death of 1 in 4 men and 1 in 5 women (more than one billion people) diagnosed with hypertension worldwide. Hypertension, the prevalence which can vary from country to country, is around 30-45% of the general population, and this rate is observed to increase with age, which will continue to be an important public health problem today and in the future. Worldwide, only one out of every 5 adults (about 21%) has hypertension under control. It is seen that the risk of cardiovascular morbidity and mortality is higher in patients whose blood pressure cannot be controlled. It is important to control hypertension in order to prevent cardiovascular diseases (CVD), also patients should comply with their treatment and health recommendations.

Motivational interviewing is a client-centered communication technique that reveals the behavior change and desire for change by helping the person to understand the problem or problems arising from himself, to discover the problem, to discover and solve the ambivalence.In this study, it is thought that motivational interviews structured according to the health belief model can be effective on cardiovascular disease risks and healthy lifestyle behavior changes in patients with an essential hypertension diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* Those who are registered with any of the family physicians in the Family Health Center where the research will be conducted.
* Being in the age range of 30-59
* Having a physician-diagnosed essential hypertension
* Having estimated 10-year CHD risk ≥ 10% based on the Framingham risk score
* Being a literate

Exclusion Criteria:

* Having a disease like coronary artery disease, heart failure, angina, myocardial infarction, cerebrovascular diseases, cancer, or kidney failure.
* Having a pacemaker
* Having a disease like chronic obstructive pulmonary disease, neurological disorder, or psychosis and schizophrenia with severe mental illness
* Has a learning disability or communication disability
* Being pregnant
* Being morbid obese (BMI ≥50 kg/m2)

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — In order for the assignments to the study and control groups to be made equally and homogeneously, 80 people in the study group will be determined by using the "stratified randomization" method, one of the randomization subgroups, according to the baseline risk factors in a balanced way in terms of the gender variable, which is one of the prognostic factors.
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic and Diastolic Blood Pressure at 3 months | 3rd month
  Systolic and diastolic blood pressure
Change from Baseline Systolic and Diastolic Blood Pressure at 6 months | 6th month
  Systolic and diastolic blood pressure
Change from Baseline 10-year and 30-year Framingham Cardiovascular Risk Score at 3 months | 3rd month
  The risk of developing cardiovascular disease in both the next 10 and 30 years will be calculated using the "Framingham cardiovascular risk score". According to the Framingham cardiovascular risk score, individuals with an estimated 10-year cardiovascular heart disease risk of <10% are considered low-risk, those between 10% and 20% are considered intermediate-risk, and individuals ≥20% are considered high-risk. The 30-year risk score estimates the 'overall' CVD risk with scores ranging from 0% to 100%. Persons with a 30-year risk score of < 12% are defined as low risk, between 12% and 40% as intermediate risk, and ≥ 40% as high risk.
Change from Baseline 10-year and 30-year Framingham Cardiovascular Risk Score at 6 months | 6th month
  The risk of developing cardiovascular disease in both the next 10 and 30 years will be calculated using the "Framingham cardiovascular risk score". According to the Framingham cardiovascular risk score, individuals with an estimated 10-year cardiovascular heart disease risk of <10% are considered low-risk, those between 10% and 20% are considered intermediate-risk, and individuals ≥20% are considered high-risk. The 30-year risk score estimates the 'overall' CVD risk with scores ranging from 0% to 100%. Persons with a 30-year risk score of < 12% are defined as low risk, between 12% and 40% as intermediate risk, and ≥ 40% as high risk.
Change from Baseline Healthy Lifestyle Behaviors at 6 months | 6th month
  "Healthy Lifestyle Behaviors Scale II" will be used to determine the healthy lifestyle behavior changes of the participants. A minimum of 52 and a maximum of 208 points can be obtained from the scale. Increasing scores from the scale indicate that individuals develop positive healthy lifestyle behaviors.

SECONDARY OUTCOMES:
Change from Baseline Cardiovascular Disease Risk Awareness Level at 3 months | 3rd month
  The "Cardiovascular Disease Risk Awareness Assessment Scale" will be used to evaluate the awareness of individuals with a diagnosis of essential hypertension about the risks associated with cardiovascular diseases. A minimum of 14 and a maximum of 56 points can be obtained from the scale. The higher scores obtained from the scale, the higher the awareness of cardiovascular diseases.
Change from Baseline Cardiovascular Disease Risk Awareness Level at 6 months | 6th month
  The "Cardiovascular Disease Risk Awareness Assessment Scale" will be used to evaluate the awareness of individuals with a diagnosis of essential hypertension about the risks associated with cardiovascular diseases. A minimum of 14 and a maximum of 56 points can be obtained from the scale. The higher scores obtained from the scale, the higher the awareness of cardiovascular diseases.
Change from Baseline Cardiovascular Diseases Risk Factors Knowledge Level at 3 months | 3rd month
  "Cardiovascular Diseases Risk Factors Knowledge Level" will be used to determine the knowledge level of the participants on cardiovascular disease risk factors. The highest total score that can be obtained from the scale is 28, and the higher score, the higher the level of knowledge.
Change from Baseline Cardiovascular Diseases Risk Factors Knowledge Level at 6 months | 6th month
  "Cardiovascular Diseases Risk Factors Knowledge Level" will be used to determine the knowledge level of the participants on cardiovascular disease risk factors. The highest total score that can be obtained from the scale is 28, and the higher score, the higher the level of knowledge.
Change from Baseline Motivation Level, Behavior Level and Self-efficacy Level in Hypertension Self-care at 6 months | 6th month
  The "Hypertension Self-Care Profile" will be used to evaluate the behavior change, motivation, and confidence levels of the participants in hypertension self-care related to lifestyle changes, and drug compliance. The hypertension self-care profile has three sub-dimensions: "Behavior", "Motivation" and "Self-efficacy". Each of the three sub-dimensions is scored separately, resulting in scores ranging from 20 to 80. Increased scores from the scale represent better self-care for a patient with hypertension.
Change from Baseline Compliance Level for Hypertension Treatment at 6 months | 6th month
  "Hill-Bone Compliance to High Blood Pressure Therapy Scale" will be used to evaluate the compliance level of the participants to hypertension treatment. A minimum score of 0 and a maximum score of 42 can be obtained from the scale, and a score of 0 indicates perfect compliance with treatment. A high total score on the scale indicates a decrease in compliance with treatment.
Change from Baseline Physical Activity Level at 6 months | 6th month
  "Physical Activity Questionnaire for Primary Care" will be used to evaluate the physical activity levels of the participants. The scale is applied to individuals between the ages of 16-74 and gives results at four levels: active, moderately active, less active and inactive.
Change from Baseline Life Quality at 6 months | 6th month
  "SF-12 Quality of Life Scale" will be used to evaluate the quality of life of the participants. Both the physical component summary score and the mental component summary score range from 0-to 100. A higher score is indicative of better health.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Duru, PhD, Principal Investigator — Department of Public Health Nursing, Eskisehir Osmangazi University, Turkey
Locations (1):
- Işıklar Family Health Center, Eskişehir, Tepebaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No